CLINICAL TRIAL: NCT01208636
Title: Environmental & Genetic Influences on Vitamin D Status
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Laura Armas, Creighton University
Other Study IDs: Creighton9
Record Dates: First submitted 2010-08-30; First posted 2010-09-24 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D deficiency; Sun; Genetics
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood was obtained for genetic testing of selected 13 candidate genes important for vitamin D metabolism
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sun exposed people: Sun exposure >3 hours daily for at least 5 days weekly for the last 3 months.

SUMMARY:
The purpose of this study is to determine the effect of environmental and genetic influences on Vitamin D status.

DETAILED DESCRIPTION:
Vitamin D deficiency is a common problem. The principal source of vitamin D for humans is solar exposure, with cutaneous synthesis of vitamin D by photoconversion of 7-dehydrocholesterol in the skin to pre-vitamin D3. Latitude, altitude, season, skin pigmentation, and age are recognized factors that influence how much vitamin D can be made by solar exposure. Surprisingly, Vitamin D deficiency has been described in people dwelling in southern Florida and in surfers in Hawaii. We hypothesize that genetic variations in vitamin metabolism accounts for these differences.

ELIGIBILITY:
Inclusion Criteria:

* Able to consent and come for a study visit.
* Male or female between ages 18-60.
* Sun exposure >3 hours daily for at least 5 days weekly for the last 3 months.

Exclusion Criteria:

* Unable to consent or come to a visit
* Taking Vitamin D supplements, anticonvulsants, barbiturates, steroids, having granulomatous disease, or liver or kidney disease as these medications and conditions interfere with Vitamin D metabolism.
* Related to another participant by blood.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will include 50 "healthy" unrelated community dwelling males or females.
  The subjects will be between ages 18-60.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
25(OH)D levels | 1 month
  25(OH)D levels were measured at the only visit

SECONDARY OUTCOMES:
Genetic testing of 13 candidate genes | 1 month
  13 candidate genes were tested and their relationship to 25(OH)D examined.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Armas, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States